CLINICAL TRIAL: NCT04623281
Title: Haemodialysis Outcomes & Patient Empowerment Study 02
Acronym: HOPE-02
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other); patientMpower Ltd. (Industry); Design to Value Ltd (Unknown); Enterprise Ireland (Other Government)
Responsible Party: Sponsor
Other Study IDs: HOPE-02
Record Dates: First submitted 2020-10-23; First posted 2020-11-10 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-10

CONDITIONS: End Stage Renal Disease; Dialysis; Complications; Volume Overload
Keywords: Sensor; Volume Overload; Dialysis; Bioimpedance
MeSH Terms: conditions — Kidney Failure, Chronic; Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Observational group of 10 haemodialysis patients following usual care for 3 weeks.
  Interventions: Device: Sixty device

INTERVENTIONS:
Device: Sixty device — Prototype wearable hydration monitor to be worn by patient during dialysis and at night

SUMMARY:
Pilot-scale, single-arm,observational study to assess the utility and acceptability of a wearable hydration monitor in haemodialysis patients compared with bioimpedance and haemodialysis machine data.

DETAILED DESCRIPTION:
Pilot-scale, single-arm,observational study to assess the utility and acceptability of a wearable hydration monitor in haemodialysis patients compared with bioimpedance and haemodialysis machine data.

The Sixty device uses diffuse reflectance spectroscopy to measure fluid status.

20 patients will be assessed during the study observation period.

10 patients undergo an observation period of approximately three weeks. The patients will be asked to wear the Sixty device during dialysis and at night throughout the study observation period.

Following the completion of this 3 week observation period, an additional 10 patients will wear the Sixty device as per the protocol for 3 weeks.

Haemodialysis parameters will be assessed as usual during the study.

Bioimpedance measurements will be taken pre and post-dialysis once weekly during the mid-week dialysis session:

Patient-reported symptoms related to haemodialysis will be recorded, including symptoms of hypervolaemia and hypovolaemia.

ELIGIBILITY:
Inclusion Criteria:

* On haemodialysis in an ambulatory care setting.
* Demonstrates understanding of correct use of the Sixty device.
* Capable and willing to measure blood pressure at home on a daily basis.
* Willing to give written informed consent.

Exclusion Criteria:

* Conditions precluding use of bioimpedance (e.g. Implantable Cardioverter Defibrillator, pacemakers, hearing aids, pregnancy).
* Significant confusion or any concomitant medical condition, which would limit the ability of the patient to record symptoms or other parameters.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Require maintenance haemodialysis in an ambulatory care setting. Study will be conducted in a single centre in a tertiary hospital. Patients with a range of baseline fluid statuses will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of Sixty device versus bioimpedance | 3 weeks
  The primary endpoint will be to evaluate the accuracy of the Sixty device data in assessing volume in haemodialysis patients compared to bioimpedance
  Bioimpedance measurements will be performed using the Fresenius Body Composition Monitor (BCM)

SECONDARY OUTCOMES:
Comparison of changes in volume status as determined by Sixty device versus fluid removed per unit of time during haemodialysis session | 3 weeks
  Fluid removed (mls/ unit of time)
Comparison of changes in volume status as determined by Sixty device versus blood pressure | 3 weeks
  Blood pressure (mmHg)
Comparison of changes in volume status as determined by Sixty device versus change in weight pre and post dialysis | 3 weeks
  Weight (kg)
Comparison of changes in volume status as determined by Sixty device versus change in blood volume monitoring | 3 weeks
  Blood volume monitoring: Relative blood volume (%)
Acceptability of Sixty device | 3 weeks
  The patient's opinion of the acceptability of the Sixty device as assessed by their response to a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Renal Dialysis Centre, Beaumont Hospital, Principal Investigator — RCSI
Locations (1):
- Beaumont Hospital, Dublin, Leinster, Ireland

REFERENCES:
- [Derived] Sandys V, Edwards C, McAleese P, O'Hare E, O'Seaghdha C. Protocol of a pilot-scale, single-arm, observational study to assess the utility and acceptability of a wearable hydration monitor in haemodialysis patients. Pilot Feasibility Stud. 2022 Jan 24;8(1):17. doi: 10.1186/s40814-022-00976-7. PMID 35073985

DOCUMENTS (1):
  • Study Protocol (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04623281/Prot_000.pdf